CLINICAL TRIAL: NCT02916433
Title: Octreotide for Management of Bronchorrhea in Mechanically Ventilated Patients: A Randomized Controlled Trial
Brief Title: Octreotide for Management of Bronchorrhea in Mechanically Ventilated Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danbury Hospital (Other)
Responsible Party: Principal Investigator, Joann Petrini, PhD, MPH, Director, Clinical Outcomes and Health Services Research, Danbury Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1101
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Octreotide; Sputum
MeSH Terms: interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): This group will continue to receive treatments that have already been initiated to manage bronchial secretions.
- Octreotide (Experimental): This group will continue to receive treatments that have already been initiated to manage bronchial secretions. Additionally, this group will receive parenteral octreotide.
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Octreotide
  Other Names: Sandostatin; Sandostatin LAR
  Arms: Octreotide

SUMMARY:
The purpose of this study is to determine whether administration of octreotide (12-25 mcg/hour) for 72 hours in combination with the standard of care treatment is effective in reducing bronchorrhea (excessive airway secretions) in mechanically ventilated patients. The use of this drug (octreotide) to manage bronchorrhea has not been approved by the United States Food and Drug Administration (FDA) and is used as an experimental drug in this research study. We are anticipating to enroll approximately 30 subjects in this study at Danbury Hospital, with 15 patients randomly assigned to the "Routine Care" group, which will serve as the control group, and 15 patients randomly assigned to the octreotide group. Control group will only receive the standard of care and will not receive this drug. Total subject participation in this study will be for 4 days (96 hours) or until their breathing tube is removed (extubation), whichever occurs first.

DETAILED DESCRIPTION:
Octreotide is widely available and has a relatively low cost (about $17/day in our hospital). In the United States, it has been used widely in outpatient and inpatient settings for over 16 years, mostly for various endocrinopathies and gastrointestinal variceal bleeds but also for a number of other pathologies. It is considered by clinicians to be an overall well-tolerated medication, with fewer significant side-effects compared to systemic steroids and scopolamine. If octreotide is proven to be an effective mucoregulator, it may become an essential tool used in the intensive care units throughout the world.

The purpose of this study is to evaluate effectiveness of including parenteral octreotide (12-25 mcg/hour for 72 hours) in addition to the other standard of care treatments deemed necessary by the ICU attending physician in managing bronchorrhea in mechanically ventilated patients. It is hypothesized that octreotide decreases excessive bronchial secretions and shortens time to extubation.

This study is an open-label, randomized controlled trial. Patients will be randomized into two groups of 15, "Routine Care" group, which will serve as the control group, and "Octreotide" group. The amount of bronchial secretions is routinely measured in all mechanically ventilated patients. Once the Primary Team identifies a patient as a candidate for the study (based on the inclusion and exclusion criteria) and an informed consent has been obtained, the baseline volume of bronchial secretions per 12-hour period will be recorded and a security envelope containing group assignment will be opened by the ICU attending. Both groups will continue to receive treatments that have already been initiated to manage bronchial secretions. In addition, "Octreotide" group will receive parenteral octreotide, while "Routine Care" group will receive care as deemed necessary by the Primary Team. The rate of bronchial secretions will be measured and recorded daily; the changes, relative to the baseline measurements, will be compared between the groups. These interventions will be continued for 72 hours or until extubation or withdrawal from the study, whichever occurs earlier. Subsequently, the standard of care management, as determined by the Primary Team, will be resumed.

Primary outcome: Change in the rate of bronchial secretion, as compared to the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients are being weaned from mechanical ventilation
* Excessive bronchial secretions (over 200 ml/24 hours) is deemed by the Primary Team to be a major barrier to extubation

Exclusion Criteria:

* Known hypersensitivity to octreotide
* Persistent bradycardia (HR < 60)
* Mobitz type II or 3rd degree heart block in patients without a pacemaker
* Patients being treated with intravenous agents for hypertensive urgency or emergency
* Surgical patients
* Initiation of therapy with systemic or inhaled steroids within 72 hours prior to the enrollment into the study, as these may further change the rate of secretions*
* Initiation of therapy with systemic or inhaled anticholinergics within 48 hours prior to the enrollment into the study, as these may further change the rate of secretions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhijith Hegde, MD, Principal Investigator — Danbury Hospital
Locations (1):
- Danbury Hospital, Danbury, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Octreotide: This group will continue to receive treatments that have already been initiated to manage bronchial secretions. Additionally, this group will receive parenteral octreotide.
  Octreotide
Period: Overall Study
Arm/Group | Usual Care | Octreotide
Started | 3 | 2
Completed | 1 | 2
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Octreotide | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (NA) — the standard deviation is a measure of the amount of variation and here we have data from only one participant | 59.5 (2.1) | 61 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Bronchial Secretion Volume Over Preceding 24 Hour Period
Description: Change in the rate of bronchial secretion at 24, 48, and 72 hours post-intervention initiation, as compared to the baseline rate
Time Frame: baseline, 24, 48, 72 hours
Measure: Number; unit: mL/24 hr
Groups:
- Usual Care: This patient have received treatments that have already been initiated to manage bronchial secretions. Below are the bronchial secretion rate at 24, 48, 72 hours.
- Octreotide #1; Octreotide #2: This patient have received treatments that have already been initiated to manage bronchial secretions. Additionally, this patient received parenteral octreotide. Below are the bronchial secretion rate at 24, 48, 72 hours.
Arm/Group | Usual Care | Octreotide #1 | Octreotide #2
Number analyzed (Participants) | 1 | 1 | 1
mL/24 hr
  Baseline | 220 | 310 | 200
  24 hr time point | 70 | 185 | 185
  48 hr time point | 195 | 120 | 170
  72 hr time point | 25 | NA — Patient discharged before this time point | 140

2. Secondary Outcome: Extubation Within 72 Hours
Description: Percentage of patients who were extubated within 72 hours of intervention initiation
Time Frame: 72 hours
Measure: Number; unit: percentage of patients
Arm/Group | Usual Care | Octreotide
Number analyzed (Participants) | 1 | 2
percentage of patients | 0 | 50

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each subject from the time informed consent was signed until termination from the study, up to 72 hours per subject
Arm/Group | Usual Care | Octreotide
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
Investigators were only able to enroll 5 patients in 2 years, therefore, study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT02916433/Prot_SAP_000.pdf